CLINICAL TRIAL: NCT02181270
Title: Attenuation of Interhepatic Fat and Hepatic Biomarkers With Exercise
Brief Title: Changes in Intrahepatic Lipids With Exercise
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Missouri-Columbia (Other)
Responsible Party: Principal Investigator, Jill Kanaley, professor, University of Missouri-Columbia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: IHEEX
Record Dates: First submitted 2014-06-30; First posted 2014-07-03 (Estimated); Last update posted 2018-01-23 (Actual); Status verified 2018-01

CONDITIONS: Obese
Keywords: NAFLD; obesity; ck18; blood lipids; high intensity exercise training; individuals; >5% liver fat
MeSH Terms: conditions — Obesity; Non-alcoholic Fatty Liver Disease | interventions — High-Intensity Interval Training

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- high intensity exercise (Experimental): High-intensity interval exercise (HIIE): Subjects will perform 5-10 minute warm-up (50% VO2peak). Subjects will then exercise at an exercise intensity that corresponds to 90% HRmax, for 4 minutes. This will be followed by 3 min of exercise at 55% HRmax. Four of these exercise intervals/recovery periods will be completed. The total exercise commitment will be ~45 minutes
  Interventions: Other: high intensity exercise
- Continuous moderate exercise group (Experimental): Continuous moderate exercise group (CME): Subjects will perform a 5-10 minute warm-up at 50% VO2peak. Thereafter, the intensity of exercise will be increased to 70% VO2peak by increasing the speed and incline of the treadmill. Subjects will exercise at this intensity for 60 minutes.
  Interventions: Other: continuous moderate exercise

INTERVENTIONS:
Other: high intensity exercise — Subjects will perform 5-10 minute warm-up (50% VO2peak). Subjects will then exercise at an exercise intensity that corresponds to 90% HRmax, for 4 minutes. This will be followed by 3 min of exercise at 55% HRmax. Four of these exercise intervals/recovery periods will be completed. The total exercise commitment will be ~45 minutes
  Arms: high intensity exercise
Other: continuous moderate exercise — Subjects will perform a 5-10 minute warm-up at 50% VO2peak. Thereafter, the intensity of exercise will be increased to 70% VO2peak by increasing the speed and incline of the treadmill. Subjects will exercise at this intensity for 60 minutes.
  Arms: Continuous moderate exercise group

SUMMARY:
Individuals with obesity and particular type 2 diabetes have abnormally high levels of fat in liver cells and are at increased risk for cardiovascular and liver-related mortality. Prior research has shown that caloric restriction, exercise, and behavior modification can help lower hepatic fat levels in these individuals. Additional research has also shown that exercise independent of weight loss can reduce hepatic fat content in obese humans. The current exercise guidelines do not specify what type or what intensity of exercise is required to induce such reductions in hepatic fat. Thus, the purpose for doing this study is to determine if there are differential effects on liver fat with 4 wk of high intensity intermittent exercise compared with continuous moderate exercise in obese individuals.

DETAILED DESCRIPTION:
Subjects will complete a liver spectroscopy scan to ensure that they have 5% body fat. Subjects passing screening will then have body composition measurement and aerobic capacity (VO2 peak) measured. Blood samples will also be taken and subjects will complete an oral glucose tolerance test. Upon completion of this testing subjects will be randomized into one of two groups: Continuous moderate exercise group or High-intensity interval exercise .

Continuous moderate exercise group (CME): Subjects will perform a 5-10 minute warm-up at 50% VO2peak. Thereafter, the intensity of exercise will be increased to 70% VO2peak by increasing the speed and incline of the treadmill. Subjects will exercise at this intensity for 60 minutes. A 5 minute cool-down (50% VO2peak).

High-intensity interval exercise (HIIE): Subjects will perform 5-10 minute warm-up (50% VO2peak). Following the warm-up, the speed and incline of the treadmill will be increased so that subjects reach an exercise intensity that corresponds to 90% Heart Rate max. Subjects will exercise at this intensity for 4 minutes, after which the treadmill speed and incline will be reduced to an intensity between 55% and 70% Heart Rate max for 3 minutes. This procedure will be replicated three additional times for a total of four intervals/recovery periods. The total exercise commitment will be ~45 minutes.

After 4 wk of exercise training all subjects will undergo all of the initial testing.

ELIGIBILITY:
Inclusion Criteria:

* Overweight or obese with a body mass index between 30-45 kg/m2.
* No known cardiovascular, kidney, or liver disease.
* No extreme hypertension (>160 mm Hg systolic and/or > 100 mm Hg diastolic).
* Not being treated with exogenous insulin.
* No history of surgery for weight loss and weight stable for prior 3 months (weight change < 3 kg).
* Non-exerciser (< 20 minutes of exercise 2 days per week).
* Between 21-60 yr of age

Exclusion Criteria:

* History of alcohol use (> 20 g/day for males and > 10 g/day for females)
* Kidney or liver disease.
* Extreme hypertension >160 mm Hg systolic and/or > 100 mm Hg diastolic.
* Waist measurement greater than 60"
* Magnetic Resonance Spectroscopy scan with less than 5% of liver fat
* A history of surgery for weight loss.
* Exerciser (>20 minutes of exercise at least 2 days per week)
* Pregnant or lactating
* <21 or >60 yr of age

Ages: 21 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 57 (Actual)
Dates: Start 2013-10 (Actual); Primary Completion 2017-06-01 (Actual); Study Completion 2017-06-01 (Actual)

PRIMARY OUTCOMES:
percent of intrahepatic fat as measured by magnetic resonance spectroscopy | 6 weeks

SECONDARY OUTCOMES:
plasma cytokeratin 18 (ck18) units: (U/I) | 6 weeks

OTHER OUTCOMES:
blood measures of blood lipids (triglycerides, cholesterol, high density lipoproteins (HDL) ) | 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Jill Kanaley, PhD, Principal Investigator — University of Missouri-Columbia
Locations (1):
- University of Missouri, Columbia, Missouri, United States

REFERENCES:
- [Derived] Winn NC, Liu Y, Rector RS, Parks EJ, Ibdah JA, Kanaley JA. Energy-matched moderate and high intensity exercise training improves nonalcoholic fatty liver disease risk independent of changes in body mass or abdominal adiposity - A randomized trial. Metabolism. 2018 Jan;78:128-140. doi: 10.1016/j.metabol.2017.08.012. Epub 2017 Sep 20. PMID 28941598